CLINICAL TRIAL: NCT01459133
Title: Single Site, Single Subject, Treatment IND With Mannkind Corporation's Technosphere
Brief Title: Single Site, Single Subject, Treatment IND With Mannkind Corporation's Technosphere Inhalation System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to register Treatment IND with the US Food And Drug Administration's new process of establishing TLS encryption for email correspondence.
Sponsor: South Orange County Endocrinology (Other)
Collaborators: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND110021
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes
Keywords: investigational; inhaled insulin product
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Technosphere® Insulin Inhalation System (Experimental): Single Site, Single Subject use of Technosphere® Insulin Inhalation System
  Interventions: Drug: Technosphere® Insulin Inhalation System

INTERVENTIONS:
Drug: Technosphere® Insulin Inhalation System — Single Site, Single Subject use of Technosphere® Insulin Inhalation System

SUMMARY:
The purpose of this program is to allow patients with diabetes and with specific medical needs which require them to use this investigational inhaled insulin product in order to adequately manage their diabetes. Treatment use of this investigational product is only anticipated when exceptional need is identified by a treating physician on a per patient case by case review.

DETAILED DESCRIPTION:
This program is for patients who have been diagnosed with diabetes mellitus and has established a need for treatment with this investigational product documented by a health care professional. The treating doctor, or a member of his/her staff, will discuss the specific requirements for participation with the subject.

INVESTIGATIONAL PRODUCT DESCRIPTION:

Technosphere® Insulin Inhalation System includes Technosphere® Insulin Inhalation Powder and inhaler. The Inhalation Powder comes in 10 unit and 20 unit cartridges.

ELIGIBILITY:
Inclusion Criteria:

Documented diagnosis with diabetes mellitus and have established a need for treatment with the investigational product.

Local Ethics Committee approval has been documented, as needed. Patient has signed the Informed Consent Form for participation. Patient has successfully completed training on the Technosphere Insulin Inhalation System.

Exclusion Criteria:

Allergy to Insulin. Smoking in the previous 6-months. History of asthma or COPD or any other significant pulmonary disease, or exposure to pulmonary toxins.

Clinical significant abnormality in screening laboratory tests. Positive pregnancy test or the intention to become pregnant. Women of childbearing age without appropriate method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Inhaled Insulin versus Subcutaneous Insulin in a patient who receives inadequate response from subcutaneous alone. | 12-months
  Evaluate fasting plasma glucose and hemoglobin a1c

CONTACTS AND LOCATIONS:
Locations (1):
- South Orange County Endocrinology, Laguna Hills, California, United States